CLINICAL TRIAL: NCT00004581
Title: A Randomized, Open-Label, Phase III Study of ABT-378/Ritonavir in Combination With Nevirapine and Two Nucleoside Reverse Transcriptase Inhibitors (NRTIs) vs. Investigator Selected Protease Inhibitor(s) in Combination With Nevirapine and Two NRTIs in Antiretroviral-Experienced HIV-Infected Subjects
Brief Title: A Study to Compare Two Anti-HIV Drug Combinations in HIV-Infected Patients Who Have Previously Received Anti-HIV Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Purpose: Treatment
Other Study IDs: 285D; M98-888
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Nevirapine; HIV Protease Inhibitors; Ritonavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; ABT 378
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Nevirapine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Nevirapine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of 2 anti-HIV drug combinations in HIV-infected patients. Both combinations will include nevirapine (NVP), 2 nucleoside reverse transcriptase inhibitors (NRTIs), and at least 1 protease inhibitor (PI). One combination will include a new protease inhibitor, ABT-378, combined in a capsule with ritonavir (RTV).

DETAILED DESCRIPTION:
Patients receive 1 of the following:

1. ABT-378/RTV plus NVP plus 2 NRTIs; or
2. Investigator-selected PI(s) plus NVP plus 2 NRTIs.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 12 years old.
* Are HIV-positive and have a viral load (level of HIV in the blood) of 1,000 - 100,000 copies/ml.
* Are currently taking an anti-HIV drug combination that includes 1 PI and 2 NRTIs, and that has not been changed in at least 12 weeks.
* Are naive to (have never taken) at least 1 NRTI, other than zalcitabine or abacavir.
* Agree to abstinence or use of an effective barrier method (e.g., condom) of birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have an active illness.
* Have received treatment for any active opportunistic (AIDS-related) infection within 30 days of study entry.
* Have ever received a nonnucleoside reverse transcriptase inhibitor (NNRTI).
* Have received investigational (not yet approved by the FDA) drugs within 30 days of study entry.
* Have received treatment with a PI other than their current PI.
* Are receiving chemotherapy for cancer.
* Are pregnant or breast-feeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Locations (88):
- United States (46):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Body Positive, Phoenix, Arizona
  - Pacific Oaks Med Group, Beverly Hills, California
  - Orange County Ctr for Special Immunology, Fountain Valley, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Tower ID Med Associates, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Yale Univ / AIDS Clinical Trials Unit, New Haven, Connecticut
  - Univ of Miami School of Medicine, Miami, Florida
  - Infectious Disease Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Emory Univ, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Tulane Univ Med School, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Boston Med Ctr, Boston, Massachusetts
  - Community Research Initiative of New England, Brookline, Massachusetts
  - Univ of Michigan Hospitals and Health Ctrs, Ann Arbor, Michigan
  - Abbott Northwestern Hosp, Minneapolis, Minnesota
  - Saint Michael's Med Ctr / Dept of Infectious Diseases, Newark, New Jersey
  - St Michaels Med Ctr, Newark, New Jersey
  - Beth Israel Med Ctr, New York, New York
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Howard Grossman, New York, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - SUNY at Stony Brook / Div of Infectious Disease, Stony Brook, New York
  - Duke Univ Med Ctr / Infectious Disease Clinic, Durham, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - Oregon Health Sciences Univ, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Stephen Hauptman, Philadelphia, Pennsylvania
  - The Miriam Hosp, Providence, Rhode Island
  - Oaklawn Physicians Group, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Univ of Texas / Med Branch at Galveston, Galveston, Texas
  - Joseph C Gathe, Houston, Texas
  - Univ of Utah Med School / Clinical Trials Ctr, Salt Lake City, Utah
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Univ of Virginia Health Sciences Ctr, Charlottesville, Virginia
  - Univ of Wisconsin, Madison, Wisconsin
- Royal Brisbane Hosp, Herston, Australia
- Pulmologisches Zentrum Der Stadt Wien, Vienna, Austria
- Brazil (5):
  - Hosp Evandro Chagas Fioernz, Manguinhos RJ
  - Castelo, São Paulo
  - Fundacao Zerbini Casa Da Aids, São Paulo
  - Hosp Do Servidor Publico Estadual De Sao Paulo, São Paulo
  - Hosp Heliopolis, São Paulo
- Canada (7):
  - Saint Paul's Hosp, Vancouver, British Columbia
  - Ottawa General Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Ctr, Toronto, Ontario
  - Toronto Gen Hosp, Toronto, Ontario
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Clinique Medicale L'Actuele, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
- Denmark (3):
  - Righospitalet, Copenhagen
  - Hvidovre Univ Hosp, Hvidovre
  - Odense Univ Hosp, Odense C
- France (4):
  - CHU De Bicetre, Paris
  - Groupe Hospitalier Bichat-Claude Bernard, Paris
  - Hopital Gustave Dron, Tourcoing
  - Hopital Paul Brousse, Villejuif
- Germany (6):
  - EPIMED, Berlin
  - Univ Zu Koeln, Cologne
  - Heinrich Heine Universitat, Düsseldorf
  - Klinikum Der Johann Wolfgang Goethe Universitat, Frankfurt
  - Allgemeines Krankenhaus St Georg, Hamburg
  - Aids Study Group Mannheim, Mannheim
- Ctr of AIDS Diagnosis and Treatment, Warsaw, Poland
- Ponce Univ Hosp, Ponce, Puerto Rico
- South Africa (2):
  - Miller, Belford Gardens
  - Cyrildene, Johannesburg
- Spain (6):
  - Hosp Germans Trias I Pujol, Barcelona
  - Hosp Carlos III, Madrid
  - Hosp De Mostoles, Madrid
  - Hosp Doce De Octubre, Madrid
  - Hosp La Paz, Madrid
  - Hosp Virgen Del Rocio, Seville
- Universitatsspital Zurich, Zurich, Switzerland
- United Kingdom (4):
  - Brighton Gen Hosp, Brighton
  - Chelsea and Westminster Hosp, London
  - Imperial College School of Medicine, London
  - Royal Free Hosp, London